CLINICAL TRIAL: NCT07194655
Title: Study on the Immediate Analgesic Effect of Yanglingquan Acupoint Treatment for Biliary Colic
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Tianjin Hospital of Integrated Traditional Chinese and Western Medicine (Unknown)
Responsible Party: Principal Investigator, Jiawen Dong, physiciancertified doctor, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKYY_YX_IRB_SOP_016(F）_002_04
Record Dates: First submitted 2025-09-16; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Biliary Colic
Keywords: Biliary colic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Drug therapy only
- Acupuncture group A (Experimental): Acupuncture at the Yanglingquan point
  Interventions: Other: Acupuncture at the Yanglingquan point
- Acupuncture group B (Experimental): Acupuncture at the Xiabai Point
  Interventions: Other: Acupuncture at the Xiabai Point
- Acupuncture group C (Sham Comparator): Acupuncture at non-meridian points
  Interventions: Other: Acupuncture at non-meridian points

INTERVENTIONS:
Other: Acupuncture at the Yanglingquan point — Acupuncture at the Yanglingquan point
  Arms: Acupuncture group A
Other: Acupuncture at the Xiabai Point — Acupuncture at the Xiabai Point
  Arms: Acupuncture group B
Other: Acupuncture at non-meridian points — Acupuncture at non-meridian points
  Arms: Acupuncture group C

SUMMARY:
Guided by traditional meridian and acupoint theory, conducting standardized, large-sample, multicenter randomized controlled trials (RCTs) to evaluate the clinical efficacy of pattern differentiation and meridian-based acupoint selection for biliary colic across multiple levels can provide high-quality research evidence for developing evidence-based guidelines or optimal treatment protocols. This holds significant importance for enhancing the clinical efficacy of acupuncture in treating biliary colic and promoting its widespread clinical application. Therefore, this study will conduct a multicenter, large-sample randomized controlled trial comparing the clinical effects of acupuncture at Yanglingquan (GB34) versus drug therapy for acute cholecystitis biliary colic. It aims to investigate the clinical efficacy and safety of acupuncture treatment for acute cholecystitis biliary colic.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for cholecystitis according to both Chinese and Western medicine;
* Patients exhibiting clinical manifestations of biliary colic with a Visual Analogue Scale (VAS) score >4;
* Aged 18 to 65 years;
* Patients provide informed consent and voluntarily participate in this study.

Exclusion Criteria:

* Patients meeting criteria for emergency surgery;
* Patients with psychiatric issues unable to cooperate with treatment;
* Patients with severe complications such as suppurative cholecystitis, suppurative cholangitis, acute pancreatitis, gallbladder perforation, tumors, or severe infections;
* Patients with other serious comorbidities including liver, brain, kidney, or cardiovascular diseases;
* Patients with severe local lesions (e.g., infections, burns, scalds) where acupuncture is contraindicated;
* Pregnant women and lactating women;
* Patients who have already undergone other treatment modalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the study is limited to specific, self-identified genders
Enrollment: 248 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Simplified McGill Pain Questionnaire (SF-MPQ) Score：Visual Analogue Scale (VAS) | One week from enrollment to the end of treatment
  This is a simple, single-dimensional method for measuring pain intensity, which consists of a 10-centimeter horizontal line. The left end is marked with "No pain", and the right end is marked with "most severe pain". The patient marks a point on the line representing the current intensity of their pain.The higher the score, the worse the result.
Simplified McGill Pain Questionnaire (SF-MPQ) Score：Pain Index (PRI) | One week from enrollment to the end of treatment
  It contains 15 pain description words, which are divided into two categories: sensory items (11 words) : throbbing pain, shooting pain, stabbing pain, sharp pain, spastic pain, biting pain, heat-burning pain, aching pain, heavy pain, touch pain, tearing pain. Emotional items (4 words) : Tiredness - feeling exhausted, nauseating, fear, punishment - feeling tormented. PRI scoring criteria: 0 = None; 1= mild; 2= moderate; 3= Severe. Calculate the total score. The higher the score, the worse the result.
Simplified McGill Pain Questionnaire (SF-MPQ) Score-Current Pain Intensity (PPI) | One week from enrollment to the end of treatment
  This is a single overall score for the current intensity of pain. It adopts a 5-point scoring method: 0= painless; 1= Mild pain; 2= uncomfortable pain; 3= Distress pain; 4= Terrifying pain; 5= Extreme pain. The higher the score, the worse the result.
Gallstones Traditional Chinese Medicine Syndrome Scoring | One week from enrollment to the end of treatment
  Referring to the relevant content of the "Clinical Guidelines for New Traditional Chinese Medicine Drugs (Trial)" 2002 edition "Gallstones" chapter, a quantitative scoring table for TCM syndromes was formulated. This study scored three symptoms: right upper abdominal pain, tenderness in the gallbladder area, and nausea and vomiting. The main symptoms (pain type) were scored as 0 points, 3 points, 6 points, and 9 points respectively for asymptomatic, mild symptoms, moderate symptoms, and severe symptoms. For secondary symptoms (nausea and vomiting), scores of 0, 1, 2, and 3 are given based on the above conditions. The minimum value is 0 points and the maximum value is 12 points.The scoring time is before treatment and 12 hours after treatment.The higher the score, the worse the result.

SECONDARY OUTCOMES:
Biliary tract ultrasound | One week from enrollment to the end of treatment
  Maximum longitudinal diameter (L) and anterior-posterior diameter (W) of the gallbladder
The levels of plasma C-reactive protein (CRP) | One week from enrollment to the end of treatment
  The levels of plasma C-reactive protein (CRP)were detected before the start of treatment and 30 minutes after treatment.The measurement unit is mg/L.
The levels of plasma cholecystokinin (CCK) | One week from enrollment to the end of treatment
  The levels of plasma cholecystokinin (CCK) were detected before the start of treatment and 30 minutes after treatment.The measurement unit is pmol/L.
The levels of plasma β -endorphin (β-EP) | One week from enrollment to the end of treatment
  The levels of plasma β -endorphin (β-EP) were detected before the start of treatment and 30 minutes after treatment.The measurement unit is pg/mL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Begona Barroso M, de Jong AP. A new design for large, dilute sample loading in capillary electrophoresis. J Capillary Electrophor. 1998 Jan-Apr;5(1-2):1-7. PMID 10327363
- [Background] Patel R, Tse JR, Shen L, Bingham DB, Kamaya A. Improving Diagnosis of Acute Cholecystitis with US: New Paradigms. Radiographics. 2024 Dec;44(12):e240032. doi: 10.1148/rg.240032. PMID 39541246